CLINICAL TRIAL: NCT00149097
Title: Autonomic Nervous System Activity in the Pathogenesis of the Lipodystrophy Syndrome in HIV-Infected Patients.
Brief Title: Role of the Autonomic Nervous System in HIV-Lipodystrophy
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Hector-Stiftung (Other)
Responsible Party: Prof. Georg Behrens, Hannover Medical School
Other Study IDs: ANS-M26
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections; Lipodystrophy-Syndrome
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to characterise the influence of the autonomic nervous system activity on the development of the lipodystrophy syndrome in HIV-infected patients by measuring heart rate variability and various metabolic pathways in HIV patients receiving highly active antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Age above 18 years
* No AIDS defining event during last 6 months
* No infection during last 6 weeks
* No concommitant drug interfering with insulin sensitivity and ANS-activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed HIV infection and no active opportunistic infection during the last 2 months.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2005-03; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg MN Behrens, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Fliers E, Sauerwein HP, Romijn JA, Reiss P, van der Valk M, Kalsbeek A, Kreier F, Buijs RM. HIV-associated adipose redistribution syndrome as a selective autonomic neuropathy. Lancet. 2003 Nov 22;362(9397):1758-60. doi: 10.1016/s0140-6736(03)14858-1. PMID 14643128